CLINICAL TRIAL: NCT01727869
Title: Study of REGN1400 Alone and in Combination With Erlotinib or Cetuximab in Patients With Certain Types of Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R1400-ST-1113
Record Dates: First submitted 2012-11-02; First posted 2012-11-16 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Erlotinib Hydrochloride; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Dosing regimen 1: REGN1400 or REGN1400 and erlotinib or REGN1400 and cetuximab
  Interventions: Drug: REGN1400; Drug: Erlotinib; Drug: Cetuximab
- Cohort 2 (Experimental): Dosing regimen 2: REGN1400 or REGN1400 and erlotinib or REGN1400 and cetuximab
  Interventions: Drug: REGN1400; Drug: Erlotinib; Drug: Cetuximab
- Cohort 3 (Experimental): Dosing regimen 3: REGN1400 or REGN1400 and erlotinib or REGN1400 and cetuximab
  Interventions: Drug: REGN1400; Drug: Erlotinib; Drug: Cetuximab

INTERVENTIONS:
Drug: REGN1400
Drug: Erlotinib
Drug: Cetuximab

SUMMARY:
This is an open-label, multicenter, ascending multiple dose study of REGN1400 alone and in combination with erlotinib or cetuximab administered to patients with certain types of cancer.

ELIGIBILITY:
Inclusion Criteria include, but are not limited to, the following:

1. Confirmed diagnosis of certain unresectable or metastatic cancers
2. Adequate Eastern Cooperative Oncology Group (ECOG) performance status
3. Adequate hepatic, renal and bone marrow function
4. Resolution of toxicity from prior therapy to grade less than/ = to 1

Exclusion Criteria include, but are not limited to, the following:

1. Active brain metastases
2. Thromboembolic events < 6 months prior to study
3. Patients with a recent history (within 5 years) of another malignancy.
4. Investigational or any antitumor treatment with a maximum of 4 half-lives or administered 30 days prior to the initial administration of REGN1400
5. Patients who are pregnant or nursing
6. Prior treatment with ErbB3 inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to characterize the safety profile of REGN1400 alone and in combination with erlotinib or cetuximab | Day 1 - Day 28
  Safety will be assessed through analysis of laboratory data, physical examination findings and vital signs according to the schedule of assessments, in addition to the spontaneous reporting of adverse events according to CTCAE version 4.

SECONDARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | Day 1 to Day 28
  Determine a recommended phase 2 dose (RP2D) of REGN1400 in combination with erlotinib or cetuximab

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (6):
- United States (6):
  - Santa Monica, California
  - Atlanta, Georgia
  - Detroit, Michigan
  - Buffalo, New York
  - New York, New York
  - San Antonio, Texas